CLINICAL TRIAL: NCT00502281
Title: Timed Intercourse Versus Intrauterine Insemination in Infertile Patients Undergoing Gonadotropin Ovarian Stimulation
Brief Title: Controlled Ovarian Stimulation Followed by Timed Intercourse or Intrauterine Insemination in Infertile PCOS Patients
Status: Suspended | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, Associate Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/2006e
Record Dates: First submitted 2007-07-12; First posted 2007-07-17 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Gonadotropins; Infertility; Intrauterine insemination; PCOS; Timed intercourse; Treatment
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility

ARMS (2):
- Group A (Active Comparator): COS followed by TI
  Interventions: Drug: highly purified urinary FSH; Behavioral: timed intercourses, intrauterine insemination
- Group B (Active Comparator): COS followed by IUI
  Interventions: Drug: highly purified urinary FSH; Behavioral: timed intercourses, intrauterine insemination

INTERVENTIONS:
Drug: highly purified urinary FSH
Behavioral: timed intercourses, intrauterine insemination

SUMMARY:
At the present the first options to induce ovulation in polycystic ovary syndrome with anovulatory infertility are clomiphene citrate (CC) and metformin. Notwithstanding the effectiveness of CC and metformin alone or in a sequential or combined regimen, a percentage of patients ranging from 5% to 30% remain anovulatory. For these patients, the use of gonadotropins for controlled ovarian stimulation (COS) is indicated.

Moreover, to date it isn't clear if COS should be followed by timed intercourse (TI) or intrauterine insemination (IUI).

The aim of the present study will be to compare TI and IUI in infertile PCOS patients undergoing COS in terms of cost-benefit.

DETAILED DESCRIPTION:
Infertile PCOS patients who remain anovulatory after CC or metformin treatment will be enrolled. All patients will receive gonadotropins in low-dose step-up protocol for COS, and randomized to receive three trials of TI (group A) or IUI (group B).

All patients eligible will undergo baseline assessment consisting of anthropometric, hormonal, and ultrasonographic evaluations.

In all patients the COS will be obtained using highly purified urinary FSH in a low-dose step-up protocol, and both TI and IUI will be performed after 35 hours from ovulation induction with human chorionic gonadotropin.

During the study, the clinical and reproductive outcomes, the adverse experience will be evaluated in each patient.

Data will be analyzed using the intention-to-treat principle and a P value of 0.05 or less will be considered significant. Continuous variables will be analyzed with the unpaired t test and general linear model for repeated measures analysis with Bonferroni test for the post-hoc analysis as required. For categorical variables, the Pearson chi-square and Fisher's exact tests will be used. Cumulative pregnancy rate, our primary end-point, will be calculated by the Kaplan-Maier method, and the differences between the two groups will be assessed with the log-rank test. Cox proportional-hazards model will be used to calculate the hazard ratio for new pregnancy in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome (using NIH criteria)
* Anovulatory infertility (using WHO criteria)

Exclusion Criteria:

* Age <18 or >35 years
* Severe obesity (BMI >35)
* Neoplastic, metabolic, hepatic, and cardiovascular disorders or other concurrent medical illnesses
* Hypothyroidism, hyperprolactinemia, Cushing's syndrome, and non-classical congenital adrenal hyperplasia
* Current or previous (within the last six months) use of oral contraceptives, glucocorticoids, antiandrogens, anti-obesity drugs, hormonal drugs
* Intention to start a diet or a specific program of physical activity
* Organic pelvic diseases
* Previous pelvic surgery
* Suspected peritoneal factor infertility
* Tubal or male factor infertility or sub-fertility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-01; Primary Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 3 months

SECONDARY OUTCOMES:
Abortion rate | 3 months
Adverse events | 3 months
OHSS | 3 months
Multiple pregnancy rate | 3 months
Costs | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Department of Obstetrics & Gynecology, University "Magna Graecia" of Catanzaro; Francesco Orio, MD, Principal Investigator — Department of Endocrinology, University "Federico II" of Naples; Achille Tolino, MD, Principal Investigator — Department of Obstetrics & Gynecology, University "Federico II" of Naples
Locations (1):
- Pugliese Hospital, Catanzaro, Catanzaro, CZ, Italy